CLINICAL TRIAL: NCT02426216
Title: Molecular Effects of a Multi-carotenoids (MCS) New Agent on Prostate Cancer Chemoprevention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 201412038RINB
Record Dates: First submitted 2015-04-09; First posted 2015-04-24 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; chemoprevention; biomarker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, prostate tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Group A: Subjects who fullfil all eligibility criteria of the MCS-8 protocol and consent to enroll the study.
- Group B: Group B: Subjects who fullfil the definition of elevated risk for prostate cancer by the MCS-8 protocol but did not sign up for the MCS-8 study.

SUMMARY:
This is to prospectively investigate whether the chemopreventive agent, MCS, may favorably alter biomarker expression, whether serum carotenoids levels are associated with biomarkers levels, and whether the alterations of biomarker expression may reflect the cancer risk as shown by cancer incidence at the end of the clinical trial.

DETAILED DESCRIPTION:
Many epidemiological studies have shown that nutrients or elements from tomato or other plants, including lycopene and multi-carotenoids, may reduce the risk of prostate cancer, especially those of lethal cancer. Studies have also shown that multi-carotenoids may reduce serum PSA levels in prostate cancer patients. MCS is a patented, multi-carotenoids-rich, purely botanic agent. The investigators' previous Phase II and III clinical trials (US FDA and TFDA, 600 subjects, studies finished, data in analysis) have shown that there were no MCS-related serious adverse events (SAE). MCS may relieve urinary symptoms in men with BPH and PSA was reduced in men with elevated PSA. So, the investigators are initiating a large multi-center phase II randomized study (MCS-8, N=702) in Taiwan, to study if MCS can reduce the risk of prostate cancer. High risk patients will be assigned to take oral daily 30, 15, and 0 (placebo) mg of MCS (1:1:1). The investigators will compare the cumulative prostate cancer incidence among groups and the change from baseline in serum carotenoids levels.

(MCS-8-TWN-II Clinicaltrials.gov NCT02042807)

ELIGIBILITY:
Inclusion criteria:

1. Subject of MCS-8 study inclusion criteria of MCS-8 study

1. high-risk subjects of prostate cancer.
2. Male subject with age from 50 to 75 years old.
3. No active urinary tract infection (UTI) or bacterial prostatitis.
4. Subject is able to understand and willing to comply with the study procedures and has signed the informed consent form (ICF).

exclusion criteria of MCS-8 study

1. Subjects' elevated PSA is deemed by the investigators solely to inflammation or infection of the prostate.
2. Subjects who are or will be taking long-term hormonal agents that may affect the normal physiology of sex hormone function.
3. Subjects with a PSA > 10.0 ng/ml.
4. Subjects with a history of prostate cancer.
5. Subjects are currently taking or planning to take oral bile acid sequestrants.
6. Subjects have malabsorption conditions.
7. Subject participated in another investigational agent study in the past 30 days or is planning to do so during the study period.
8. Subjects are considered ineligible for the study as judged by the investigator.
9. Other malignancies except non-melanoma skin cancer.

2. Subject is eligible for MCS-8 study but did not sign up for the MCS-8 study.

Exclusion criteria:

Subject is not able to understand and willing to comply with the study procedures and has not signed the informed consent form (ICF).

Note: (MCS-8-TWN-II Clinicaltrials.gov NCT02042807)

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are increased risk of prostate cancer
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative histologically proven prostate cancer | up to 104 weeks
  Cumulative histologically proven prostate cancer incidence at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan